CLINICAL TRIAL: NCT01061606
Title: Pilot Phase II Study of Temsirolimus in Patients With Recurrent Mixed Mesodermal and Mullerian Tumors (Carcinosarcoma) of the Uterus
Brief Title: Temsirolimus in Treating Patients With Recurrent or Persistent Cancer of the Uterus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02989; NCI-2012-02989 (Other: CTRP (Clinical Trial Reporting Program)); 8167 (Other: CTEP); N01CM00038 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-09

CONDITIONS: Recurrent Uterine Sarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel

SUMMARY:
This phase II trial is studying how well temsirolimus works in treating patients with recurrent or persistent cancer of the uterus. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the efficacy of Temsirolimus in women with recurrent or persistent (after primary therapy) Carcinosarcoma (MMMT) of the uterus.

II. Assess the safety and tolerability of Temsirolimus in this patient population.

III. Evaluate secondary efficacy endpoints of time to tumor progression, progression-free survival (PFS), 6 month PFS rate, and duration of response.

SECONDARY OBJECTIVES:

I. Overall survival II.Duration of Response III. Time to progression IV. Time to treatment failure

OUTLINE: This is a multicenter study.

Patients receive temsirolimus IV over 30 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Carcinosarcoma (MMMT)
* Measurable disease;
* Only one prior systemic treatments after primary adjuvant treatment for persistent or metastatic disease are permitted,
* Radiation therapy (adjuvant or palliative) must be completed ≥ 4 weeks prior to registration
* Required laboratory values obtained =< 7 days prior to registration:
* Absolute Neutrophil Count (ANC) >= 1500/mm^3
* Platelets >= 75,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Direct bilirubin =< 1.5 x upper limit of normal (ULN)
* Alkaline phosphatase =< 2.5 x ULN (≤ 5 x ULN if liver metastasis is present)
* SGOT(AST) =< 2.5 x ULN (≤ 5 x ULN if liver metastasis is present)
* Creatinine =< 1.5 x ULN
* Fasting serum cholesterol ≤ 350mg/dL (9.0 mmol/L)
* Triglycerides ≤ 1.5 x ULN

  * Patients with Triglyceride levels > 1.5 x ULN can be started on lipid lowering agents and reevaluated within 1 week; if levels go to ≤ 1.5 x ULN, they can be considered for the trial and continue the lipid lowering agents
* International Normalized Ratio (INR) ≤ 1.5 (unless the patient is on full dose warfarin)
* ECOG Performance Status (PS) 0-1
* Capable of understanding the investigational nature, potential risks and benefits of the study and able to provide valid informed consent
* Full-dose anticoagulants, if a patient is receiving full-dose anticoagulants, the following criteria should be met for enrollment:

  * The subject must have an in-range INR (usually between 2 and 3) on a stable dose of warfarin or on stable dose of LMW heparin
* Patients who have had prior anthracycline must have a normal ejection fraction on LVEF assessment by MUGA or Echo ≤ 4 weeks prior to registration
* Availability of tissue samples or blocks (from the primary tumor or metastases) for tumor studies
* Willingness to donate blood for correlative marker studies

Exclusion Criteria:

* Prior therapy with Temsirolimus or another mTOR inhibitors
* Patients cannot be receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) nor any other CYP3A4 inducer such as rifampin or St. John's wort
* Untreated central nervous system (CNS) metastases; exceptions: patients with known CNS metastases can be enrolled if the brain metastases have been adequately treated and there is no evidence of progression or hemorrhage after treatment as ascertained by clinical examination and brain imaging (MRI or CT) ≤ 12 weeks prior to registration and no ongoing requirement for steroids

  * Anticonvulsants (stable dose) are allowed
  * Patients who had surgical resection of CNS metastases or brain biopsy ≤ 3 months prior to registration will be excluded
* Pregnant or lactating wome
* Currently active, second malignancy other than non-melanoma skin cancers; - Other uncontrolled serious medical or psychiatric condition (e.g. cardiac arrhythmias, diabetes, etc.)
* Active infection requiring antibiotics
* Received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of endometrial cancer
* Radiation therapy to > 50% of marrow bearing areas

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Einstein, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (20):
- United States (20):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope, Duarte, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - City of Hope Medical Group Inc, Pasadena, California
  - University of California at Davis Cancer Center, Sacramento, California
  - University of Connecticut, Farmington, Connecticut
  - Yale University, New Haven, Connecticut
  - Morristown Memorial Hospital, Morristown, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Women's Cancer Care Associates LLC, Albany, New York
  - Beth Israel Medical Center, New York, New York
  - New York University Langone Medical Center, New York, New York
  - Saint Luke's Roosevelt Hospital Center - Roosevelt Division, New York, New York
  - Presbyterian-Weill Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Children's Hospital of New York Presbyterian, New York, New York
  - Columbia University College of Physicians and Surgeons, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 patients were enrolled at two institutions between July 2010 and January 2012
Period: Overall Study
Arm/Group | Treatment (Temsirolimus)
Started | 8
Completed | 0
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Disease Progression | 4
Not completed — alternative therapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3
  Black | 2
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate, in Terms of the Proportion of Confirmed Tumor Responses (CR or PR) Assessed Using RECIST
Time Frame: Up to 3 years
Measure: Number; unit: participants
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 6
participants
  Disease progression | 4
  Stable disease | 2

2. Primary Outcome: Progression Free Survival
Description: The 6-month progression-free rate is defined as the total number of efficacy-evaluable patients on study without documentation of disease progression 6 months from registration divided by the total number of efficacy-evaluable patients enrolled on study.
Time Frame: 6 months from registration
Population: The study concluded terminated early and patients were not followed.
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Time to event distributions will be estimated using the Kaplan-Meier method.
Time Frame: From registration to death, assessed up to 3 years
Population: The study concluded terminated early and patients were not followed.
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response, Defined for All Evaluable Patients Who Have Achieved an Objective Response as the Date at Which the Patient's Objective Status is First Noted to be Either a CR or PR to the Date Progression is Documented
Description: Median duration of response and the confidence interval for the median duration will be computed.
Time Frame: Up to 3 years
Population: The study concluded terminated early and patients were not followed.
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure will be evaluated using the method of Kaplan-Meier.
Time Frame: From study registration to the date patients end treatment, assessed up to 3 years
Population: The study concluded terminated early and patients were not followed.
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Progression
Time Frame: Time to progression is defined as the time from registration to disease progression.
Population: The study concluded terminated early and patients were not followed.
Arm/Group | Treatment (Temsirolimus)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Temsirolimus)
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Temsirolimus) (N=8)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Urinary Tract infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Death NOS (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Temsirolimus) (N=8)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left eye twitching (Eye disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Rasch: acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Mucositis: oral (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Euphoria (Psychiatric disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less